CLINICAL TRIAL: NCT07177339
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Study of the Efficacy and Safety of Early Depemokimab Initiation as add-on Treatment in COPD Patients With Type 2 Inflammation
Brief Title: eValuating the Efficacy and Safety of InitiatinG depemokImab earLy therApy iN Chronic Obstructive Pulmonary Disorder (COPD) With Type 2 Inflammation
Acronym: VIGILANT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 224295; 2025-521108-23 (Other: EU CT Number)
Record Dates: First submitted 2025-09-15; First posted 2025-09-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Depemokimab; Chronic Obstructive Pulmonary Disorder; COPD; Type 2 inflammation; Eosinophilic phenotype; Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a double-blind study in which participants care providers investigators and outcome assessors will be blinded to the study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Depemokimab (Experimental): Participants with Chronic Obstructive Pulmonary Disorder (COPD) with Type 2 inflammation will receive Depemokimab in combination with existing Standard of Care (SoC).
  Interventions: Drug: Depemokimab
- Placebo (Experimental): Participants with COPD with Type 2 inflammation will receive matching Placebo in combination with existing SoC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Depemokimab — Depemokimab will be administered.
  Arms: Depemokimab
Drug: Placebo — Matching placebo will be administered.
  Arms: Placebo

SUMMARY:
Depemokimab is being developed as a treatment for individuals with moderate to severe Chronic Obstructive Pulmonary Disorder (COPD). The aim of this study is to assess the efficacy and safety of early initiation of depemokimab as an add-on medicine in participants with moderate to severe COPD with type 2 inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Male or eligible female participants
* Eosinophilic phenotype measured using Blood Eosinophil Count (BEC)
* Moderate to severe COPD, defined as

  * A clinically documented history of COPD for at least 1 year
  * A post-salbutamol Forced expiratory volume in one second (FEV1)/Forced vital capacity (FVC) ratio of less than (<)0.70 and a post-salbutamol FEV1 greater than (>)30 percent (%) and <80% predicted normal values
* Elevated risk for exacerbations, defined as

  * A well-documented history of only 1 moderate COPD exacerbation in the prior 12 months and
  * The presence of risk factors for future exacerbations/deterioration such as:
  * Modified Medical Research Council (mMRC) dyspnea score >= 2
  * COPD Assessment Test (CAT) >= 15
  * Post-bronchodilator FEV1 < 50% predicted
  * Chronic bronchitis
* Smoking status: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years at Screening.
* Dual (Inhaled corticosteroid (ICS)+ Long-acting beta2-adrenergic receptor agonist [LABA] or LABA+ Long-acting muscarinic receptor antagonist [LAMA]) or triple (ICS+LABA+LAMA) inhaler therapy as assessed by the investigator for at least 3 months
* Body mass index (BMI) >=16 kilograms per square meter (kg/m^2)

Exclusion Criteria:

* The Investigator must judge that COPD is the primary diagnosis accounting for the clinical manifestations of lung disease, and clinical manifestations of lung disease where primary diagnosis is not COPD are excluded

  * Participants with a current or prior physician diagnosis of asthma
  * Participants with childhood asthma are permitted, provided that childhood asthma has resolved before 18 years of age and has not recurred
* Other clinically significant lung disease: The Investigator must judge that COPD is the primary diagnosis accounting for the clinical manifestations of the lung disease.
* COPD severity: Participants with more than one moderate exacerbation or severe exacerbation in the past 12 months prior to Visit 1
* COPD stability: Participants with pneumonia, COPD exacerbation, or lower respiratory tract infection within the 4 weeks prior to Visit 1
* Lung resection: Participants with a history of, or plan for lung volume reduction surgery/endobronchial valve procedure
* Pulmonary rehabilitation: Participants in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1
* Chronic hypercapnia requiring non-invasive positive pressure ventilation (NIPPV) use including Bi-Level Positive Airway Pressure (BiPAP) or Continuous Positive Airway Pressure (CPAP) are excluded
* Continuous oxygen: Participants requiring oxygen supplementation for COPD

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1196 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2029-11-02 (Estimated); Study Completion 2029-12-14 (Estimated)

PRIMARY OUTCOMES:
Annualized Rate of Moderate/Severe Exacerbations | From Baseline Up to Week 156
  Moderate exacerbations are defined as clinically significant exacerbations that require treatment with oral/systemic corticosteroids and/or antibiotics. Severe exacerbations are defined as clinically significant exacerbations that require in-patient hospitalization (that is greater than or equal to [>=] 24 hours) or result in death. The frequency of moderate/ severe exacerbations expressed as an annualized rate of moderate or severe exacerbations will be reported.

SECONDARY OUTCOMES:
Time to First Moderate/Severe Exacerbation | From Baseline Up to Week 156
  Moderate exacerbations are defined as clinically significant exacerbations that require treatment with oral/systemic corticosteroids and/or antibiotics. Severe exacerbations are defined as clinically significant exacerbations that require in-patient hospitalization (that is greater than or equal to (>=) 24 hours) or result in death.
Change from Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score at Week 52 | From Baseline up to Week 52
  The SGRQ total score will be measured using the SGRQ for COPD [SGRQ-C]. The SGRQ-C is a 40-item participant questionnaire designed to measure health impairment by addressing the frequency of respiratory symptoms (questions 1-7) and the participants current state (questions 8-14). The questions are designed to be completed by the participant. The total score will be calculated on 0-100 rating scale and scores expressed as a percentage of overall impairment. Higher scores indicate greater impairment of health.
Change from Baseline in Evaluating Respiratory Symptoms (E-RS): COPD Total Score at Week 52 | From Baseline up to Week 52
  E-RS: COPD consists of 11 items from the 14-item Exacerbations of Chronic Pulmonary Disease Tool - Patient Reported Outcomes (EXACT) instrument. E-RS: COPD is intended to capture information related to the respiratory symptoms of COPD, that is, breathlessness, cough, sputum production, chest congestion, and chest tightness. The E-RS: COPD has a scoring range of 0 to 40, higher scores indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- GSK Investigational Site, Doral, Florida, United States
- China (5):
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Guilin
  - GSK Investigational Site, Jiangmen
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Taizhou

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf